CLINICAL TRIAL: NCT03428854
Title: Adenomyosis: Genomic Mechanisms and Biological Response
Status: Withdrawn | Type: Observational
Why Stopped: The study never got funded so never started enrolling
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Kho, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: 0000
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Adenomyosis; Abnormal Uterine Bleeding
MeSH Terms: conditions — Adenomyosis; Metrorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: LNG-IUS — Levnorgestrel containing IUD
  Other Names: Mirena

SUMMARY:
Examination of genomic and biologic responses to LNG-IUS in patients with adenomyosis.

DETAILED DESCRIPTION:
Examination of genomic and biologic responses to LNG-IUS in patients with adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal bleeding in the presence of Adenomyosis as demonstrated by MRI

Exclusion Criteria:

* Other causes of abnormal bleeding such as fibroids, endometrial polyps, malignancy
* Presence of endometriosis

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Uterus required
Study Population: Women with abnormal uterine bleeding due to adenomyosis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Menstrual blood loss | 12 months
  Pictorial blood loss assessment chart

SECONDARY OUTCOMES:
Quality of Life | 12 months
  SF-12
Pain | 12 months
  Visual analog scale